CLINICAL TRIAL: NCT05011279
Title: "Sitting Less, Moving More": Designing a Digital Health Intervention for Black and African American Women Breast Cancer Survivors and Their At-risk Relatives (Phase II)
Brief Title: Move Together Boston Feasibility Pilot (Sit Less, Move More App for Black Breast Cancer Survivors & At-Risk Relatives)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: University of Massachusetts, Boston (Other); University of Rochester (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Catherine Marinac, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-104; U54CA156732 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-18 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Survivor; Breast Cancer; Fitness Trackers
Keywords: Digital Health Intervention; Breast Cancer Survivor; Breast Cancer; Garmin Activity Tracker; Move Together App; Fitness trackers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Study (Experimental): Participants in the pilot study will participate as members of family-based dyads (n=5 dyads). One member of each dyad will be a breast cancer survivor and one will be a blood relative.
  Study involves interviews, questionnaires, Use of Move Together app with Garmin activity tracker watch
  Interventions: Other: Move Together app/Garmin Activity Tracker

INTERVENTIONS:
Other: Move Together app/Garmin Activity Tracker — * The Move Together app allows users to set daily goals for increasing physical activity and decreasing sedentary time, track progress on goals, message their buddy, and access external educational infographics and other resource links.
  * Garmin activity tracker in this study is for participants to track their steps and sedentary time.

SUMMARY:
The purpose of this study is to develop and test a mobile app for Black/African American breast cancer survivors and their relatives, called Move Together, that promotes sitting less and moving more for better health.

DETAILED DESCRIPTION:
The purpose of this study is to develop and test a mobile app for Black/African American breast cancer survivors and their relatives, called Move Together, that promotes sitting less and moving more for better health.

This is a cross-sectional descriptive study using structured interviews and qualitative data analysis to develop an intervention, followed by a pilot test of the intervention with pre- /post- measures.

* In study phase 1,involved qualitative interviews with 5 community leader key informants, 9 breast cancer survivors and 6 first degree relatives of a survivor.
* This part of the research study is a Pilot Study, which means it is the first time that researchers are studying usability and acceptability of the Move Together app.

  * Participants in the pilot study will participate as members of family-based dyads (n=10 dyads). One member of each dyad will be a breast cancer survivor and one will be a blood relative
  * Study involves screening for eligibility, interviews, questionnaires, Use of Move Together app with Garmin activity tracker watch
  * Participation on the trial will be for 5 weeks
* About 20 people (10 survivors with 10 relatives) will participate in this part of the study, and a total of 58 people in the whole study.

ELIGIBILITY:
Inclusion Criteria:

* 1a) Key informants (for interviews)

  * Members of the community/advisory groups, community health centers, or faith-based network members (e.g., Pink and Black, Faces of Faith).
  * English speaking adults.
* (1b) Breast cancer survivors and relatives (for interviews)

  * Self-identify as Black or African American
  * Age 18 and over
  * English speaking
  * Female breast cancer survivor status post curative antineoplastic treatment (except ongoing hormonal treatment) with no evidence of disease, OR a first degree blood relative (parent, child, or full sibling), of any gender, of a so defined breast cancer survivor
  * Self-report ever using a smart phone
* (2) Breast cancer survivors and relatives (for user testing/interviews)

  * Self-identify as Black or African American
  * Age 18 and over
  * English speaking
  * Female breast cancer survivor status post curative antineoplastic treatment (except ongoing hormonal treatment) with no evidence of disease, OR a first degree blood relative (parent, child, or full sibling), of any gender, of a so defined breast cancer survivor
  * Self-report willing/able to download the app for testing on a smart phone
  * Self-report willing/able to meet via Zoom for interview
* (3) Breast cancer survivors and relatives/"buddies" (for pilot testing)

  * Self-identify as Black or African American
  * Age 18 and over
  * English speaking
  * Breast cancer survivor status post curative antineoplastic treatment (except ongoing hormonal treatment) with no evidence of disease, OR a blood relative, of any gender, of a so defined breast cancer survivor
  * Self-report willing/able to participate with a blood relative in survivor relative dyad
  * Self-report willing/able to download the app for use on a smart phone
  * Self-report willing/able to meet via Zoom for instructions and interview

Exclusion Criteria:

* (1a) Key informants (for interviews)

  --None
* (1b) Breast cancer survivors and relatives (for interviews)

  * Requires medically supervised physical activity (Physical Activity Readiness Question for Everyone, PAR-Q+, Question 7)
  * Pregnant women
* (2) Breast cancer survivors and relatives (for user testing/interviews)

  * Requires medically supervised physical activity (Physical Activity Readiness Question for Everyone, PAR-Q+, Question 7)
  * Pregnant women
* (3) Breast cancer survivors and relatives/"buddies" (for pilot testing)

  * Meets exclusion criterion of the Modified Physical Activity Readiness Questionnaire (PAR-Q) (modified)
  * Participated in interviews or user testing in prior phases of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Marinac, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Boston, Boston, Massachusetts
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Blazey M, Marinac C, Whiteley J, Peterson S, Burns White K, Jacques C, Lam H, Halpenny B, Patel S, Lamothe R, Wright J. Designing a Dyad-Based Digital Health Intervention to Reduce Sedentary Time in Black Breast Cancer Survivors and Their First-degree Relatives: Human-Centered Design Study. JMIR Form Res. 2023 May 24;7:e43592. doi: 10.2196/43592. PMID 37223968

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Study: Participants in the pilot study will participate as members of family-based dyads (n=5 dyads) in this single arm study. One member of each dyad will be a breast cancer survivor and one will be a blood relative.
  Study involves interviews, questionnaires, Use of Move Together app with Garmin activity tracker watch
  Move Together app/Garmin Activity Tracker: - The Move Together app allows users to set daily goals for increasing physical activity and decreasing sedentary time, track progress on goals, message their buddy, and access external educational infographics and other resource links.
  -Garmin activity tracker in this study is for participants to track their steps and sedentary time.
Period: Overall Study
Arm/Group | Pilot Study
Started | 10 (5 survivors and 5 relatives)
Completed | 10 (5 survivors and 5 relatives)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: this includes 5 survivors and 5 relatives
Groups:
- Pilot Study: Participants in the pilot study will participate as members of family-based dyads (n=5 dyads). One member of each dyad will be a breast cancer survivor and one will be a blood relative.
  Study involves interviews, questionnaires, Use of Move Together app with Garmin activity tracker watch
  Move Together app/Garmin Activity Tracker: - The Move Together app allows users to set daily goals for increasing physical activity and decreasing sedentary time, track progress on goals, message their buddy, and access external educational infographics and other resource links.
  -Garmin activity tracker in this study is for participants to track their steps and sedentary time.
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 45.9 [22 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Breast Cancer Status [Count of Participants; unit: Participants]
  Survivor | 5
  Mother of a survivor, no BRCA | 1
  Daughter of a survivor, no BRCA | 1
  Sister of a survivor, no BRCA | 2
  Niece of a survivor, no BRCA | 1

OUTCOME MEASURES:

1. Primary Outcome: System Usability Scale (SUS) Score
Description: The acceptability of the Move Together app will also be assessed with The System Usability Scale (SUS) score. The scale has 10 items. Scores range from 0-100; a SUS score above a 68 is considered above average (https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html.)
Time Frame: Assessed at 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
units on a scale | 72 (14.3)

2. Secondary Outcome: Number of Participants Screened Per Month
Description: the number of participants screened per month during recruitment period (not cumulative)
Time Frame: 4 month recruitment period
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
Participants | 5

3. Secondary Outcome: Number of Participants Enrolled Per Month
Description: number of participants consented to the study each month during enrollment period
Time Frame: 4 month enrollment period
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
Participants | 3

4. Secondary Outcome: Completion Rate
Description: number of participants who completed all aspects of the protocol
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
Participants | 10

5. Secondary Outcome: Number of Study Days
Description: number of study days in which the participants uses the Move Together app and will describe engagement with the app in a 28 day period (i.e., study days)
Time Frame: baseline to 4 weeks (28 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
days | 17.1 (8.6)

6. Secondary Outcome: Number of Participants Recruited
Description: Number of initial respondents who consent and enroll.
Time Frame: during 4 month recruitment period
Measure: Number; unit: participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
participants | 1

7. Secondary Outcome: Number of Participants Completed Study
Description: Total number of participants who completed the study
Time Frame: 4 weeks
Measure: Number; unit: number of participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
number of participants | 9

8. Secondary Outcome: Number of Participants Retained at the End of 4 Weeks
Description: Retention will be the number who remain in the study at the end of 4 weeks
Time Frame: Baseline to 4 Weeks
Measure: Number; unit: number of participants
Arm/Group | Pilot Study
Number analyzed (Participants) | 10
number of participants | 10

ADVERSE EVENTS:
Time Frame: 5 weeks
Groups:
- Single Arm of Breast Cancer Survivors (n=5) and Family Members (n=5): Participants in the single arm pilot study will participate as members of family-based dyads (n=5 dyads). One member of each dyad will be a breast cancer survivor and one will be a blood relative.
  Study involves interviews, questionnaires, Use of Move Together app with Garmin activity tracker watch
  Move Together app/Garmin Activity Tracker: - The Move Together app allows users to set daily goals for increasing physical activity and decreasing sedentary time, track progress on goals, message their buddy, and access external educational infographics and other resource links.
  -Garmin activity tracker in this study is for participants to track their steps and sedentary time.
Arm/Group | Single Arm of Breast Cancer Survivors (n=5) and Family Members (n=5)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT05011279/Prot_SAP_000.pdf